CLINICAL TRIAL: NCT03399812
Title: The Effect of Breakfast on Energy Metabolism, Appetite, and Food Intake in Men
Brief Title: Breakfast and Metabolism in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jamie Baum, Assistant Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1708038914
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Aging
MeSH Terms: interventions — Plant Proteins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey protein isolate (Experimental)
  Interventions: Dietary Supplement: Animal protein
- Pea protein isolate (Active Comparator)
  Interventions: Dietary Supplement: Plant protein

INTERVENTIONS:
Dietary Supplement: Animal protein — The animal protein intervention is a smoothie containing 40 grams of whey protein isolate.
  Arms: Whey protein isolate
Dietary Supplement: Plant protein — The animal protein intervention is a smoothie containing 40 grams of pea protein isolate.
  Arms: Pea protein isolate

SUMMARY:
This study will determine the short-term postprandial effects of protein source at breakfast on energy metabolism, markers of metabolic health, appetite, and food intake and young and older men.

ELIGIBILITY:
Inclusion Criteria:

* Male
* No medication
* Athlete (elite or professional)

Exclusion Criteria:

* Diet-related conditions
* Food allergies
* Does not regularly consume protein supplements
* Claustrophobic
* Underweight

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | Time frame is every 30 minutes for four hours following intervention.
  Energy expended per minute will be measured using indirect calorimetry.
Appetite | Time frame is every 30 minutes for four hours following intervention.
  Appetite will be assessed using a traditional 100-mm visual analog scale (VAS) (3) with opposing anchors (e.g., "extremely hungry" or "not hungry at all") at time points 15, 30, 60, 90, 120, 180 and 240 min. Questions consisted of: "how hungry do you feel at this moment", "how full do you feel at this moment", "how strong is your desire to eat this moment" and "how much food do you think you can eat at this moment." Participants were asked to place an "X" on the 100-mm VAS in the place that pertained to their perceived appetite feelings at each time point." Participants were asked to place an "X" on the 100-mm VAS in the place that pertained to their perceived appetite feelings at each time point. The averages for each time point are taken to represent the feeling of appetitive at a particular time point.

SECONDARY OUTCOMES:
24-hour food intake | Food intake will be recorded for one day.
  Food intake following the intervention will be recorded using food records.

OTHER OUTCOMES:
Appetite biomarkers | Time frame is every 30 minutes for four hours following intervention.
  PYY, CCK and orexin will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Baum, Principal Investigator — University of Arkansas, Fayetteville
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hawley AL, Gbur E, Tacinelli AM, Walker S, Murphy A, Burgess R, Baum JI. The Short-Term Effect of Whey Compared with Pea Protein on Appetite, Food Intake, and Energy Expenditure in Young and Older Men. Curr Dev Nutr. 2020 Jan 22;4(2):nzaa009. doi: 10.1093/cdn/nzaa009. eCollection 2020 Feb. PMID 32072131